CLINICAL TRIAL: NCT03988647
Title: A Phase 2 Study of Palliative Radiation Therapy and Anti-PD-1/PD-L1 Checkpoint Blockade in Patients With Metastatic Merkel Cell Carcinoma
Brief Title: Palliative RT & Anti-PD-1/PD-L1 Checkpoint Blockade in Metastatic Merkel Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Susan Pillsbury, Associate Professor of Radiation Oncology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-50888; IRB-50888 (Other: Stanford-IRB); SKIN0047 (Other: OnCore)
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Merkel Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + Palliative Radiation Therapy (Experimental): Pembrolizumab will be administered at 200 mg IV every 3 weeks as standard of care. Palliative radiation therapy will be given between the first and second cycles of immunotherapy
  Interventions: Drug: Pembrolizumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administered at 200 mg IV every 3 weeks
  Other Names: Keytruda
Radiation: Radiation Therapy — 9 Gy X 3 (27 Gy in 3 fractions), or 4-6 Gy X 5 (20-30 Gy in 5 fractions).

SUMMARY:
The primary objectives of this study are to assess 1) the safety and 2) efficacy of combining Anti-PD-1/PD-L1 blockade with palliative radiation therapy in patients with Stage IV Merkel Cell Carcinoma.

DETAILED DESCRIPTION:
The hypothesis for this study is that local radiation therapy (RT) can be safely used in combination with PD-1/PD-L1 blockade. This combination therapy may have the potential to enhance the induction of systemic anti-Merkel cell carcinoma immune responses, which will inhibit growth and kill Merkel cell tumor cells in sites of established metastases outside of the local radiation therapy field.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic Merkel Cell Carcinoma.
* Patients are eligible if they have received no more than 3 prior systemic treatments, inclusive of systemic adjuvant therapy. This includes previously untreated patients.
* Subjects with brain metastases and/or carcinomatous meningitis are eligible providing they are neurologically stable (if systemic steroids are required, subjects should be stable on the lowest clinically effective dose, as steroids may interfere with the activity of immunotherapy if administered at the time of the first Anti-PD-1/PD-L1 dose.)
* Availability of tumor tissue (fresh or archival) for central pathology review.
* Must be at least 14 days since treatment with chemotherapy, biochemotherapy, surgery, or immunotherapy, and recovered (baseline or residual Grade 1 toxicity) from any clinically significant toxicity experienced during treatment before the first dose of pembrolizumab therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of ≥ 16 weeks.
* Subjects must have measurable disease according to RECIST v1.1, and have baseline (screening/baseline) radiographic images, (e.g. CT, Positron emission tomography (PET)/CT or MRI brain, chest, abdomen, pelvis, to be determined by the attending physician) within 4 weeks of confirmation of eligibility and within 6 weeks before the initiation of pembrolizumab therapy.
* Required values for initial laboratory tests:
* White blood cells (WBC): ≥ 2000/µL (~ 2 x 109/L)
* Absolute Neutrophil Count (ANC): ≥ 1000/µL (~ 1 x 109/L) Platelets: ≥ 50 x 103/µL (~ 50 x 109/L)
* Hemoglobin: ≥ 8 g/dL
* Calculated creatinine clearance greater than 30 mL/min
* Aspartate transaminase(AST)/alanine transaminase (ALT): Less than 2.5 x upper limit of normal (ULN) for subjects without liver metastasis, less than 5 times ULN for liver metastases
* Bilirubin: less than 3.0 x ULN (except for subjects with Gilbert's Syndrome, who must have a total bilirubin of less than 3.0 mg/dL)
* Non-clinically significant laboratory abnormalities such as lipase elevation would not be an exclusion.
* No known active or chronic infection with HIV, Hepatitis B, or Hepatitis C, or active infection requiring systemic antibiotics. Testing for the above is not required unless clinically suspected.
* At least one measurable site of disease (≥ 10 mm as per RECIST v1.1 except for lymph nodes that must be 15 mm or greater on the short axis) outside of the planned palliative radiation therapy field.
* Require radiation therapy for palliation of symptoms or to prevent local progression of disease and associated complications and/or symptoms from metastases.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.
* WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Post-menopausal is defined as:

  * Amenorrhea ≥ 12 consecutive months without another cause, or
  * For women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
* Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 1 week prior to the start of investigational product.
* Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study and for up to 26 weeks after the last dose of investigational product.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or before investigational product administration.
* Subjects on any other systemic therapy for cancer, including any other experimental treatment within 2 weeks of scheduled first dose of pembrolizumab.
* Prior treatment with an anti-PD-1/PD-L1 antibody if treatment failure was due to AEs. If a subject was discontinued from the prior anti-PD-1/PD-L1 treatment due to an Adverse events (AE) or Serious adverse events (SAE), regardless of the type of event, that discontinuation constitutes an exclusion criterion. If AEs were serious enough to require a subject's withdrawal from prior treatment, the subject should be excluded from this study. The exception to the above are non-clinically significant immune-related laboratory abnormalities - these are not automatic exclusions - e.g. asymptomatic elevated amylase; responsiveness to steroids. In situations above - e.g. non-clinically significant immune-related laboratory abnormalities, each case will be considered individually and a decision made by the study team.
* A history of AEs with prior IL-2 or Interferon will not preclude subjects from entering the current study.
* Autoimmune disease: Poorly controlled autoimmune disease is excluded. Well controlled autoimmune disease (e.g. well controlled RA) will be assessed by the study team and a decision made regarding eligibility based on the degree of immunosuppression and severity of symptoms.
* Any subject who has a life-threatening condition that requires high-dose immunosuppressant(s). Steroid doses greater than 20 mg/day will exclude the patient from participation in the trial.
* Presence of known hepatitis B or hepatitis C infection, regardless of control on antiviral therapy.
* Subjects who have another active, concurrent, malignant disease are not eligible, with the exception of subjects with adequately treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or other cancers that are in remission/not measurable. Patients will be excluded if they have any known additional malignancy that requires active treatment while on treatment for Merkel Cell Carcinoma.
* Bilirubin/total bilirubin 3 or more X ULN unless conjugated bilirubin is less than or equal to the ULN.
* Evidence of symptomatic interstitial lung disease or symptomatic active, noninfectious pneumonitis.
* Participants with impaired cardiac function or clinically significant cardiac disease such as unstable angina/uncompensated heart failure, uncontrolled symptomatic arrhythmia.
* Active autoimmune disease requiring systemic T-cell immunosuppression.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment. This exclusion does not include prophylactic antibiotics or topical antibiotics.
* Known hypersensitivity to another monoclonal antibody, which cannot be controlled with standard measures (e.g. antihistamines and corticosteroids).
* Any condition that would, in the investigator's judgment, interfere with full participation in the study.
* Prior immune related AEs not meeting the conditions above.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects with acute or poorly controlled psychiatric illness or subjects who are compulsorily detained for physical (e.g., infectious disease) illness, with the exception of patients that are well supported and able to participate (e.g. paraplegia from a motor vehicle accident).
* Any underlying medical or psychiatric condition that, in the opinion of the investigator, could make the administration of anti-PD-1/PD-L1 hazardous or could obscure the interpretation of adverse events.
* Any live vaccine therapy for up to 4 weeks before or after any dose of immunotherapy on this trial.
* Any investigational agents within 2 weeks of scheduled first dose of pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Knox, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab + Palliative Radiation Therapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Palliative Radiation Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Tumor Response at both irradiated & unirradiated sites will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Basic RECIST response will be assessed by the criterion below.
  * Complete Response (CR) = Disappearance of all target lesions.
  * Partial Response (PR) = ≥0% decrease in the sum of the longest diameter (LD) of target lesions.
  * Stable disease (SD) = Small changes that do not meet any of the above criteria.
  RECIST v1.1 immune-related response will be assessed by the criterion below.
  * Immune-related CR (irCR) = Disappearance of all target lesions. Lymph nodes <10 mm in short axis.
  * Immune-related PR (irPR) = ≥30% decrease in the sum of the LD of target lesions.
  * Immune-related SD (irSD) = Failure to meet criteria for irCR or irPR in the absence of irPR.
  The outcome is reported as the number of lesions with each of the different levels of clinical response, a number without dispersion.
Time Frame: 15 months
Population: Note that basic clinical response and immune-related clinical response are distinct assessments, and each are reported for the participant.
Measure: Number; unit: tumor lesions
Arm/Group | Pembrolizumab + Palliative Radiation Therapy
Number analyzed (Participants) | 1
tumor lesions
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable disease (SD) | 1
  Immune-related complete response (irCR) | 0
  Immune-related partial response (irPR) | 0
  Immune-related stable disease (irSD) | 1

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was assessed as the duration of time from study entry to time of death or the date of last contact. The outcome is reported as OS in months.
Time Frame: 18 months
Measure: Number; unit: months
Arm/Group | Pembrolizumab + Palliative Radiation Therapy
Number analyzed (Participants) | 1
months | 18

3. Secondary Outcome: Duration of Response (DOR)
Description: The duration of response (DoR) is measured from the time the criteria are met for CR or PR (whichever is first recorded) until the date that recurrent or progressive disease is documented. Tumor response at both irradiated & unirradiated sites will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Basic RECIST response will be assessed by the criterion below.
  * CR = Disappearance of all target lesions.
  * PR = ≥0% decrease in the sum of the longest diameter (LD) of target lesions.
  * SD = Small changes that do not meet any of the above criteria.
  RECIST immune-related response will be assessed by the criterion below.
  * irCR = Disappearance of all target lesions. Lymph nodes <10 mm in short axis.
  * irPR = ≥30% decrease in the sum of the LD of target lesions.
  * irSD = Failure to meet criteria for irCR or irPR in the absence of irPR. The outcome is reported as the duration of response for each level of level of clinical response.
Time Frame: 15 months
Population: Results are reported as the duration of response for each level of tumor response.
Measure: Number; unit: months
Units Other Than Participants: lesions
Arm/Group | Pembrolizumab + Palliative Radiation Therapy
Number analyzed (Participants) | 1
Number analyzed (lesions) | 2
months
  Complete Response (CR): number analyzed (lesions) | 0
  Partial Response (PR): number analyzed (lesions) | 0
  Stable disease (SD): number analyzed (lesions) | 1
  Stable disease (SD) | 15
  Immune-related complete response: number analyzed (lesions) | 0
  Immune-related partial response (irPR): number analyzed (lesions) | 0
  Immune-related stable (irSD): number analyzed (lesions) | 1
  Immune-related stable (irSD) | 15

ADVERSE EVENTS:
Time Frame: 532 days
Arm/Group | Pembrolizumab + Palliative Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Palliative Radiation Therapy (N=1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte decreased (Investigations) | 1 (1)
Alanine transferase increase (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Back Pain (General disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03988647/Prot_SAP_000.pdf